CLINICAL TRIAL: NCT00379834
Title: 12-Month Stability of Diurnal IOP Control on Cosopt
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Anthony D. Realini, Associate Professor, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31861
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-01

CONDITIONS: Glaucoma
Keywords: glaucoma; diurnal; intraocular pressure
MeSH Terms: conditions — Glaucoma | interventions — dorzolamide-timolol combination; dorzolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cosopt (Active Comparator): Cosopt twice daily in both eyes
  Interventions: Drug: Cosopt

INTERVENTIONS:
Drug: Cosopt — Cosopt twice daily in both eyes
  Other Names: Dorzolamide/timolol fixed combination

SUMMARY:
To determine the stability of diurnal intraocular pressure in eyes with glaucoma treated with Cosopt

DETAILED DESCRIPTION:
Glaucoma is a potentially-blinding but treatable eye disease. A major risk factor for glaucoma is elevated intraocular pressure (IOP). IOP is a dynamic variable (like blood pressure)-it changes over time. The more it changes, the more likely patients are to get worse. Glaucoma is treated by lowering IOP. Cosopt is a medication that lowers IOP. Little is known about how well Cosopt reduces IOP fluctuations. In this study, we plan to measure the IOP in both eyes of 10 glaucoma patients treated with Cosopt, every 2 hours from 8am to 8pm, on five separate days over a one-year period. Untreated baseline IOP will be measured on a similar long day before beginning treatment with Cosopt. This methodology will allow us to compare IOP fluctuations with and without Cosopt, and also to learn about long-term control of IOP fluctuations in eyes treated with Cosopt.

ELIGIBILITY:
Inclusion Criteria:

* bilateral open-angle glaucoma

Exclusion Criteria:

* contraindications to Cosopt
* pathology affecting tonometry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony D Realini, MD, Principal Investigator — West Virginia University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 subjects enrolled from WVU Eye Institute between April 2006 and April 2008
Pre-assignment Details: No patients excluded at any time
Groups:
- Cosopt: Cosopt BID OU
Period: Overall Study
Arm/Group | Cosopt
Started | 10
Completed | 8
Not Completed | 2
Not completed — Time constraints | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cosopt
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Diurnal Intraocular Pressure Control
Description: Change from baseline in mean diurnal IOP (measured every two hours from 8AM to 8PM) averaged across on-treatment study visits (week 1, months 1, 6, 12)
Time Frame: 12 months
Population: Selected by level funding available
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Cosopt
Number analyzed (Participants) | 10
millimeters of mercury | -4.4 (2.0)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cosopt
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes